CLINICAL TRIAL: NCT06566131
Title: Gamified Mobile Health for Physical Activity Promotion in Autistic Adults
Brief Title: Development and Evaluation of A Game-Based Mobile App for Increasing Physical Activity in Autistic Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Autism Intervention Research Network on Physical Health (Unknown)
Responsible Party: Principal Investigator, Daehyoung Lee, PhD, Assistant Professor, University of Delaware
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2098388
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Mobile health; Gamification; Physical activity; Sedentary behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: All study participants will get the same mobile health intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PuzzleWalk (Gamified mHealth) (Experimental): PuzzleWalk integrates gamification strategies and incentivization of walking behaviors to induce target behavior changes. Capitalizing on the distinctive attributes and preferences of autistic adults, PW emphasizes the advantages of visual learning while minimizing the need for undesired face-to-face social interactions. A novel feature is its conversion algorithm that translates daily step counts into playtime for "spot the difference" puzzle games, which leverages the psychological satisfactions of autonomy, relatedness, and competence.
  Interventions: Behavioral: Gamified mobile health app

INTERVENTIONS:
Behavioral: Gamified mobile health app — Participants will receive visualized instructions about the PW use (e.g., search and download the app on App Store, navigate and understand key features, play puzzle games, and track step counts). During the 6-week intervention period, participants will receive reminders on wearing the accelerometer, using the app for potential incentives, and engaging in regular physical activities for health promotion.
  Other Names: PuzzleWalk

SUMMARY:
The clinical study aims to develop and test a gamified mobile health app called PuzzleWalk (PW) to promote physical activity (PA) and reduce sedentary behavior (SB) in autistic adults, including those with mild intellectual disabilities (ID). The study addresses the need for tailored interventions in this population, who are at higher risk for lifestyle-related chronic health conditions due to lower PA and higher SB. The upgraded version of PuzzleWalk integrates behavior change techniques and gamification strategies, such as translating step counts into puzzle game playtime, to encourage regular PA and reduce SB. The study will evaluate the app's effectiveness on preventive health behavior changes in real-world settings. The ultimate goal is to create an effective, sustainable, and scientifically validated mobile health tool to improve the health and well-being of autistic adults.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate the feasibility and acceptability of the upgraded PW in increasing PA and reducing SB in autistic adults with and without mild ID. For this field deployment study, we will employ a pre-/post-test design to examine any changes in participants' objective levels of PA and sedentary time before, during, and after the 6-week intervention. The working hypothesis is that the 6-week PW intervention will yield significant increases in accelerometer-measured daily step counts and moderate-to-vigorous PA (MVPA) (up to 5% increases from baseline) and decreases in sedentary time (up to 10% decreases from baseline). High levels of user engagement with PW app during the intervention period will be significantly associated with sustained positive behavior changes in daily step counts, MVPA, and sedentary time among participants.

We will conduct screening interviews with an emphasis on history of diagnosis and level of intellectual functioning to verify the eligibility of prospective participants. After they consent to participate in the study, we will provide them with study materials, including an accelerometer (i.e., wristwatch), a cable charger, and study instruction sheets, via shipping or in-person meetings. Prior to baseline data collection, we will use a rubric to assess participant comfort and knowledge of study procedures. After an initial 2-3-day accelerometer familiarization period, we will start the data collection, including demographics, technology and medication use, and accelerometer-derived PA and sedentary time. From week 3, participants will start to freely use the upgraded PW app after receiving visualized step-by-step user instructions and will continue to use the app until the end of week 8 (total 6-week intervention), supported by periodic reminders and reinforcement messages based on Behavior Change Techniques. PA and sedentary time measures will be collected during four time periods: Week 1 (baseline), Week 3 (intervention start), Week 5 (mid-intervention), and Week 8 (intervention end).

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 55 years
* individuals diagnosed with an autism spectrum disroder by a medical professional or self-identify as neurodivergent
* individuals who have regular access to a supported smartphone (iOS 13+ operating system)

Exclusion Criteria:

* individuals with a moderate-to-profound intellectual disability
* individuals with orthopedic conditions that significantly interfere with independent ambulation (e.g., using a wheelchair or crutches)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Changes in MVPA levels | Baseline, 3 weeks, 5 weeks, and 8 weeks
  Objective accelerometer-measured MVPA (min/day)

SECONDARY OUTCOMES:
Changes in self-reported PA | Baseline, 3 weeks, 5 weeks, and 8 weeks
  Measured using the Activities Completed over Time in 24-hours (ACT24). This is a web-based previous-day recall instrument (min/day).
Engagement with the PW app | 3 weeks, 5 weeks, and 8 weeks
  The level of user engagement in the PW app will be measured using a webmaster server that keeps track of user logs and timestamps (e.g., frequency and duration of app use and leaderboard scores). Time spent on the app in a min/day format will be calculated to represent each participant's level of user engagement.
Changes in light PA levels | Baseline, 3 weeks, 5 weeks, and 8 weeks
  Objective accelerometer-measured light PA (min/day)
Changes in steps | Baseline, 3 weeks, 5 weeks, and 8 weeks
  Objective accelerometer-measured steps (counts/day)
Changes in sedentary time | Baseline, 3 weeks, 5 weeks, and 8 weeks
  Objective accelerometer-measured sedentary time (min/day)
Changes in self-reported sedentary time | Baseline, 3 weeks, 5 weeks, and 8 weeks
  Measured using the Activities Completed over Time in 24-hours (ACT24). This is a web-based previous-day recall instrument (min/day).

CONTACTS AND LOCATIONS:
Overall Officials: Daehyoung Lee, PhD, Principal Investigator — University of Delaware
Locations (1):
- Carpenter Sports Building, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly as it will be used for refereed publications.

REFERENCES:
- [Derived] Lee D, McNulty L, Kathiravan S, Mauriello ML, Vasudevan V, Bhat A, Obrusnikova I, Suminski R. A Gamified mHealth App to Promote Physical Activity and Reduce Sedentary Behavior in Autistic Adults: Protocol for a Remotely Delivered Pilot Intervention Study. JMIR Res Protoc. 2025 Jul 22;14:e71631. doi: 10.2196/71631. PMID 40694837